CLINICAL TRIAL: NCT04757545
Title: Symptom Identification and Management in Patiens With Hematological Malignacy - A Randomized Controlled Trial Using HM-PRO
Brief Title: Symptom Identification and Management in Patients With Hematological Malignancy During Follow-up Care
Acronym: SIMPly-CARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Mary Jarden, Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: University Hospital Copenhagen
Record Dates: First submitted 2021-02-12; First posted 2021-02-17 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Hematologic Malignancy
Keywords: HM-PRO; Symptom management; Patient reported outcome
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: Two armed randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HM-PRO intervention (Active Comparator): The intervention group will have a predetermined nurseled consultation planned to assess medical status and symptom control at 0, 6 and 12 months. Seven days prior to the scheduled visit, the patient will receive an electronic invitation via RedCap to complete and send PRO data (HM-PRO). Prior to each appointment PRO data will be evaluated by a nurse from an algorithm deciding one of three tracks for the patients.
  Interventions: Other: HM-PRO
- Standard outpatient follow-up care (No Intervention): The control group will receive standard care in the outpatient clinic. The patient has a predetermined consultation appointment at the hospital one time a year with a doctor to evaluate medical status and symptom control.

INTERVENTIONS:
Other: HM-PRO — The intervention group will have a predetermined consultation appointment planned to assess medical status and symptom control. Seven days prior to the scheduled visit, the patient will receive an electronic invitation via RedCap to complete and send PRO data (HM-PRO). Prior to each appointment PRO data will be evaluated by a nurse from an algorithm deciding one of three tracks for the patients:
  1. Worsening in symptoms results in a nurse-led telephone consultation within two days guided by the symptom management manual.
  2. Minor changes in patient's symptom assessment result in a nurse-led telephone consultation within seven days using the symptom management manual.
  3. Patients that are completely stable in the symptom assessment will receive an electronic answer via min-SP (electronic patient journal) regarding the results and a new appointment, including PRO-data prior to this.
  Arms: HM-PRO intervention

SUMMARY:
The aim is to study the effect of a systematic approach to symptom identification and management with disease specific and clinically developed PRO (HM-PRO) with a 12 month follow up in outpatient care in patients with chronic hematological malignancy.

DETAILED DESCRIPTION:
Design: A two-arm prospective randomized controlled trial.

Population: Patients diagnosed with chronic myeloid leukemia (CML), clonal cytopenia of unknown significance (CCUS), myelodysplastic syndrome (MDS) or myeloproliferative neoplasia (MPN).

Patients will be recruited from the outpatient clinic at the Dept. of Hematology at Rigshospitalet in Denmark. Patients will be identified and screened by their physician. Patients who are eligible for study inclusion will hereafter be approached, informed and recruited by the primary research investigator. Included patients will be randomized and allocated 1:1 to an intervention group or a control group.

The intervention group will have a predetermined consultation appointment planned to assess medical status and symptom control. Seven days prior to the scheduled visit, the patient will receive an electronic invitation via RedCap to complete and send PRO data (HM-PRO). Prior to each appointment PRO data will be evaluated by a nurse from an algorithm deciding one of three tracks for the patients.

The control group will receive standard care in the outpatient clinic. The patient has a predetermined consultation appointment at the hospital one time a year with a doctor to evaluate medical status and symptom control.

Data Collection: The questionnaires will be distributed and completed by patients electronically via REDCap consisting of clinical data, PRO data (HM-PRO) and endpoint measures (see below).

* Primary outcome: Change in QoL measured by EORTC-QLQ-C30, global health domain, at 12 months.
* Secondary outcomes: Change in symptoms of depression and anxiety measured by HADS, change in symptom burden measured by MDASI symptom scale and clinical data outcomes at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* adults > 18 years
* diagnosed and undergoing follow up for a hematological malignancy in the outpatient clinic, Rigshospitalet
* The patients can be included approximately six months after initial diagnosis if in stable condition.
* able to manage an e-mail account

Exclusion Criteria:

* Patients who do not understand, read and speak Danish and/or have cognitive/psychiatric disorders not compatible with inclusion in a clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Change in Health related quality og life: EORTC QLQ C30 | At 12 months
  The global health domain

SECONDARY OUTCOMES:
Changes in symptoms of depression and anxiety measured by HADS | 6 and 12 months
  Hospital Anxiety and Depression score
Changes in symptom burden measured by MDASI symptom scale | 6 and 12 months
  MD Andersons Scale - core
Clinical outcomes | At baseline
  Hematological diagnosis
Patient experiences measured at PREM | 6 and 12 months
  Patient reported experience measures
Clinical outcome | Date for time of diagnosis - collected at baseline
  Time of diagnosis - date
Clinical outcome | Hospitalization during intervention period baseline - 12 months
  Frequency/dates and length of hospitalization
Clinical outcome | Number and charecter of referrals during interventions period baseline - 12 months
  Referrals to other departments and/or primary care in the municipality
Clinical outcome | From baseline - 12 months
  Add on medication
Clinical medication | Baseline
  Medication at baseline
Clinical outcome | From baseline -12 months
  Number of consultations in follow-up in dept. of hematology
Clinical outcome | Baseline, 6 and 12 months
  CPR - from laboratory test

CONTACTS AND LOCATIONS:
Overall Officials: Maja Pedersen, Ph.d. stud., Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Dept. of Hematology, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pedersen M, Larsen MT, Kornblit BT, Dahl EO, Lomborg K, Tolver A, Jarden M. Effects of nurse-led symptom management in chronic myeloid malignancies: a randomized trial. Support Care Cancer. 2025 Feb 15;33(3):196. doi: 10.1007/s00520-025-09230-1. PMID 39954038